CLINICAL TRIAL: NCT03927235
Title: The Diagnostic Yield and Safety of Transbronchial Cryobiopsy in Different Freezing Time in the Diffuse Parenchymal Lung Diseases: a Prospective Randomized Control Trial
Brief Title: The Diagnostic Yield and Safety of Transbronchial Cryobiopsy in Different Freezing Time in the Diffuse Parenchymal Lung Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Director of the Respiratory department, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-3-30
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Transbronchial Cryobiopsy; Freezing Time; Diagnostic Yield; Safety
Keywords: Transbronchial Cryobiopsy; freezing time; Diagnostic Yield; Safety; Diffuse Parenchymal Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- the freezing time of 3s (Sham Comparator): Transbronchial cryobiopsy in the freezing time of 3s
  Interventions: Procedure: Transbronchial Cryobiopsy
- the freezing time of 4s (Experimental): Transbronchial cryobiopsy in the freezing time of 4s
  Interventions: Procedure: Transbronchial Cryobiopsy
- the freezing time of 5s (Experimental): Transbronchial cryobiopsy in the freezing time of 5s
  Interventions: Procedure: Transbronchial Cryobiopsy
- the freezing time of 6s (Experimental): Transbronchial cryobiopsy in the freezing time of 6s
  Interventions: Procedure: Transbronchial Cryobiopsy

INTERVENTIONS:
Procedure: Transbronchial Cryobiopsy — Transbronchial Cryobiopsy in the Diagnosis of Diffuse Parenchymal Lung Diseases

SUMMARY:
Transbronchial cryobiopsy in different freezing time is performed in patients with undefined diffuse parenchymal lung diseases, and assess the diagnostic yield and safety.

DETAILED DESCRIPTION:
Transbronchial cryobiopsy in different freezing time is performed in patients with undefined diffuse parenchymal lung diseases, and assess the diagnostic yield and safety. This is a prospective randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

1. The patients are admitted in the institution as DPLD, while undefined after thorough history collection, laboratory examination and radiological data.
2. Transbronchial cryobiopsy(TBCB) is indicated by clinicians for definitive diagnosis and patients are content with the examination with agreement signed.
3. Blood gas analysis, routine blood test, ECG examination, coagulation function, immunological examination, chest HRCT, and liver/kidney function test have been completed.

Exclusion Criteria:

1. The radiological data indicates non-DPLD
2. The clinical examinations mentioned above are not completed.
3. The patient cannot endure or does not agree the procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-05-15 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Diagnotic yield | two weeks
  Percentage of definitive pathological diagnosis by transbronchial cryobiopsy, the alteration of original diagnosis after transbronchial cryobiopsy

SECONDARY OUTCOMES:
Complication rate | one week
  Incidence of bleeding, pneumothorax (during the procedure and within 7 days after the intervention) and exacerbations of DPLD related to the transbronchial cryobiopsy

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China